CLINICAL TRIAL: NCT01260480
Title: A Prospective, Multicenter Study, to Evaluate the Efficacy and Safety of [18F]-ML-10, a Positron Emission Tomography (PET) Imaging Radiotracer, in Early Detection of Response of Non-Hematological Tumors to Concurrent Chemoradiotherapy
Brief Title: An Efficacy and Safety Study to Assess [18F]-ML-10 in Detecting Response of Tumors to Chemotherapy and Radiation
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aposense Ltd. (Industry)
Responsible Party: Yael Cohen, Aposense
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NST-CA007
Record Dates: First submitted 2010-12-14; First posted 2010-12-15 (Estimated); Last update posted 2010-12-17 (Estimated); Status verified 2010-12

CONDITIONS: Carcinoma, Non-Small-Cell Lung; Head and Neck Neoplasms
Keywords: Carcinoma, non-small-cell lung; Head and neck neoplasms; Diagnostic imaging
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Head and Neck Neoplasms | interventions — 5-fluoropentyl-2-methylmalonic acid; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- [18F]-ML-10 (Experimental)
  Interventions: Other: [18F]-ML-10 in conjunction with PET imaging

INTERVENTIONS:
Other: [18F]-ML-10 in conjunction with PET imaging — Subjects will receive two to three intravenous (IV) doses of [18F]-ML-10. The dose for each [18F]-ML-10 dose will be 5.50 MBq/Kg or 0.15 mCi/Kg but will not exceed 500.00 MBq (13.50 mCi) per administration.

SUMMARY:
The purpose of this study is to determine whether [18F]-ML-10 used in conjunction with PET imaging is effective as an imaging tool for the early detection of response of oncological tumors in the lungs,head and neck to chemoradiation therapy.

The study will evaluate the potential of [18F]-ML-10 used in conjunction with PET imaging to distinguish early during the course of chemoradiation therapy between a tumor that responds to the therapy, and a tumor that does not respond to the therapy. Currently, this distinction is available to the physician several weeks or months after completion of therapy, using anatomical imaging (for example Computed Tomography [CT] or Magnetic Resonance Imaging [MRI]).

ELIGIBILITY:
Inclusion Criteria:

Male or female patients with either:

Newly diagnosed non small cell lung cancer (NSCLC) (Group A) who meet the following criteria:

* Previously untreated, histologically or cytologically confirmed stage IIB, IIIA or IIIB disease, without evidence of distant metastases
* A measurable primary tumor with at least one diameter > 2 cm or primary tumor extending to one or more lymph nodes which cannot be distinctively delineated as confirmed by a diagnostic quality chest CT performed within 4 weeks prior to initiation of the concurrent CRT.
* Planned to receive concurrent chemoradiotherapy as definitive treatment. The radiation dose should not exceed 70 Gy.
* Undergone the following minimum workup to confirm disease staging within 4 weeks prior to initiation of the concurrent CRT:

  * GBCA-enhanced Brain MRI or contrast enhanced CT if there are signs or symptoms suggesting brain metastases within the past 2 months.
  * If necessary to confirm stage of disease, an upper abdomen CT scan will be performed.
  * whole-body FDG PET/CT; OR
* Newly diagnosed squamous cell carcinoma of the head and neck (SCCHN) (Group B) who meet the following criteria:

  * Previously untreated, histologically or cytologically confirmed (from the primary tumor and/or lymph nodes) stage III-IV disease without evidence of distant metastases.
  * A measurable (i) primary tumor with at least one diameter ≥2 cm and (ii) lymph node with at least one diameter ≥ 2 cm as confirmed by a diagnostic quality neck CT performed within 4 weeks prior to initiation of the concurrent CRT.
  * Planned to receive concurrent chemoradiotherapy as definitive treatment. The radiation dose should not exceed 70 Gy.
  * Have undergone the following minimum workup to confirm disease staging within 4 weeks prior to initiation of the concurrent CRT:
* Whole-body FDG PET/CT.
* Patients ≥ 18 years of age.
* Able to comply with lying still during the PET/CT imaging session which may last for up to 3 hrs with intermediate breaks.
* ECOG performance status of 0, 1 or 2.
* Adequate renal function and adequate hepatic function, as assessed by standard laboratory criteria and defined as:
* Serum creatinine ≤ 1.2 times the Upper Limit of Normal (ULN).
* Total bilirubin ≤ 1.5 times the ULN.
* Asparagine aminotransferase (AST) and/or alanineaminotransferase (ALT) ≤ 2.5 times the ULN (grade 1 according to the NCI-CTCAE v.3).
* Women of child-bearing potential must have a negative blood pregnancy test at screening and use an adequate and medically acceptable contraceptive method.
* Willing and able to comply with the protocol requirements.
* Able to provide written informed consent.

Exclusion Criteria:

Exclusion criteria specific to patients with NSCLC (Group A):

* Predominant small cell carcinoma histology.
* Pure bronchioalveolar cell carcinoma histology.
* Treatment planned with chemotherapy other than a platinum-based doublet regimen.
* Malignant pleural or pericardial effusions.
* Any contraindication to perform CT with IV contrast agent.

Exclusion criteria specific to patients with SCCHN (Group B):

* Histology other than squamous cell carcinoma.
* Treatment planned with chemotherapy other than a platinum-based regimen.
* Treatment planned with cetuximab.
* Treatment with induction chemotherapy.
* Any contraindication to CT with IV contrast agent.
* Evidence of distant metastases.
* Patients who, based on the investigator's judgment, have other unstable medical conditions that may preclude safe and complete study participation.
* Treatment with any investigational drug, device or biologic agent within 30 days prior to administration of [18F]-ML-10.
* Pregnancy or lactation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2010-12; Primary Completion 2012-02 (Estimated)

PRIMARY OUTCOMES:
To characterize changes in [18F]-ML-10 uptake in the target lesion in response to chemoradiotherapy. | Between baseline and day 11 ± 1, and between baseline and day 18 ± 1

SECONDARY OUTCOMES:
To assess the correlation between the changes in the uptake of [18F]-ML-10 in the target lesion and the changes in the anatomical dimensions of the target lesion.
  To assess the correlation between the changes in the uptake of [18F]-ML-10 in the target lesion following an accumulative radiation dose of 14.4-20.0 Gy, and the changes in the anatomical dimensions of the target lesion, as assessed by the follow-up anatomical imaging by CT, performed after completion of the concurrent chemoradiotherapy (CRT).
To identify at least one parameter, derived from the changes in [18F]-ML-10 uptake that can discriminate tumors responsive to treatment from tumors that are non-responsive.
  For this parameter, various cut-off values of change will be evaluated, with corresponding estimates of sensitivity and specificity.
To perform additional analyses for all other lesions and lymph nodes with at least one diameter ≥ 2 cm treated by concurrent CRT.
To assess the safety of [18F]-ML-10 administered to cancer patients receiving concurrent CRT.

CONTACTS AND LOCATIONS:
Overall Officials: Heron Dwight, MD, Principal Investigator — University of Pittsburgh Medical Center; David Sher, MD, MPH, Principal Investigator — BWH, Harvard; Aaron Allen, MD, Study Director — Rabin Medical Center
Locations (4):
- United States (4):
  - BWH, Boston, Massachusetts
  - Holy Name Medical Center, Teaneck, New Jersey
  - Mount Sinai, New York, New York
  - University of Pittsburgh, Pittsburgh, Pennsylvania